CLINICAL TRIAL: NCT04729530
Title: The Effect of Dyson Air Purifier in Improving Asthma Control - A Randomised, Controlled Trial
Brief Title: The Effect of Dyson Air Purifier in Improving Asthma Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The David Hide Asthma & Allergy Research Centre (Other)
Collaborators: Isle of Wight NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DYSON-ASTHMA01
Record Dates: First submitted 2019-11-06; First posted 2021-01-28 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Air purifier device with standard filter cartridges installed.
  Interventions: Device: Dyson Pure Cool - Active Purifier
- Placebo (Placebo Comparator): Air purifier device with placebo (non working) filter cartridges installed.
  Interventions: Device: Dyson Pure Cool - Placebo purifier

INTERVENTIONS:
Device: Dyson Pure Cool - Active Purifier — Free standing air purifier
  Arms: Active
Device: Dyson Pure Cool - Placebo purifier — Placebo air purifier
  Arms: Placebo

SUMMARY:
To investigate the effect of reducing the level of allergens and pollutants in the bedroom and living room by placing a "Dyson air purifier", on poorly controlled asthmatic subjects.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases. Little change in morbidity and mortality has occurred despite improvements in pharmacotherapy. In the last few decades, there has been an increase in the prevalence of asthma and other allergic diseases. The precise cause for this increase in disease prevalence is not known but it has coincided with changes to the quality of indoor air with increases in the levels of allergens and pollutants. Bedroom exposure to dust-mite allergens has been linked to worsening asthma symptoms and increase in bronchial responsiveness. In places where dust mites cannot thrive, allergens from cat, cockroach and Alternaria assume importance. High indoor temperatures and humidity may, by a number of mechanisms, increase the allergenic burden, particularly the proliferation of house-dust mites and moulds. Therefore, modern living conditions are associated with a higher risk of allergen exposure causing increase in sensitisation and symptoms of asthma. In addition to allergens, the indoor environment contains other biological materials (such as microbiome and endotoxin), and pollutants (gases and particulate matter) which can adversely affect asthma development and morbidity. Indoor pollutants include smoke from cigarettes and wood, coal or gas fires, particulate materials associated with bio-fuel combustion, chemical vapours and gases including nitrogen dioxide (NO2), formaldehyde and volatile organic compounds (VOCs). The latter may come from sources including building products, cleaning agents, and paints. One such VOC is formaldehyde, which can be irritant to both upper and lower respiratory tract. Small particulate matter (PM2.5) is particularly damaging as it gets to the small airways of the lung. Major indoor sources of NO2 and particulate matter include gas stoves and cigarette smoke but outdoor sources such as traffic and industrial pollution can also contaminate indoor environment.

It has also been suggested that exposure to pollutants can potentiate the effects of allergen. Indeed, a combination of high levels of indoor pollution and allergens is causally related to the development and severity of asthma. Allergens, microbiome and pollutants can interact with each other to augment the immune response leading to harmful effects on the airways.

Thus, indoor air pollution is a significant environmental trigger for acute exacerbation of asthma (and other respiratory conditions such as COPD), leading to increasing symptoms, emergency department visits, hospital admissions and even mortality. An estimated 75% of hospital admissions for asthma are avoidable. Maintaining high air quality with lower levels of allergens and pollutants is therefore important in improving the health of individuals with asthma and other respiratory diseases. Therefore, a feasible and practical intervention that can reduce allergen and pollutant levels in the indoor air should reduce morbidity and improve asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 75 years of age with a confirmed diagnosis of mild persistent to moderate persistent asthma (BTS steps "regular preventer therapy" to "additional add-on therapies")
* ACQ6 score >1.5.

Exclusion Criteria:

* Patients with significant chronic respiratory disease such as COPD or bronchiectasis.
* Patients with any severe disease (such as cardiovascular disease, dementia etc.), where adherence to the study protocol may cause an unjustified stress.
* Those who are being treated with allergen specific immunotherapy.
* Patients with a history of significant alcohol or drug abuse.
* Patients who are taking an investigational drug for asthma.
* Patients who are unwilling, unlikely or unable to comply with the study protocol, as assessed by the study team members.
* Patients who are likely to be started on biological therapies for asthma (omalizumab, mepolizumab, reslizumab, dupilumab) during the study period.
* Pregnancy.
* Patients already using air purifiers in their dwellings.
* Patients planning to move house during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Change in asthma quality of life score | 18 months
  Change in Juniper asthma specific quality of life (AQLQ) scores: A change in score of 0.5 on the 7-point scale is considered clinically important (Minimal Important Difference).
Change in asthma control score | 18 months
  Change in asthma control composite scores using Juniper asthma control questionnaire (ACQ6). A change in score of 0.5 on the 6-point scale is considered clinically important.

SECONDARY OUTCOMES:
Change in airway responsiveness | 18 months
  Change in airway responsiveness from baseline will be compared in the two groups (as assessed by methacholine bronchial challenge).
Change in indoor pollutant level | 18 months
  Changes in indoor levels of pollutants that are recorded by Dyson purifier.
Pulmonary function: forced expiratory volume in one second (FEV1) | 18 months
  Pulmonary function as assessed by changes in forced expiratory volume in one second (FEV1),
Pulmonary function: FEV1 (forced expiratory volume in one second) /FVC (Forced Vital Capacity) ratio | 18 months
  Pulmonary function as assessed by changes FEV1/FVC (Forced Vital Capacity) ratio
Pulmonary function: mid-expiratory flows. | 18 months
  Pulmonary function as assessed by changes in mid expiratory flows.
Exhaled Nitric Oxide | 18 months
  Change in exhaled nitric oxide levels (as an indicator of airway inflammation) from baseline will be compared in the two groups.
Peak expiratory flow | 18 months
  Change in peak expiratory flow from baseline will be compared in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: S. Hasan Arshad, Principal Investigator — University of Southampton
Locations (1):
- The David Hide Asthma and Allergy Research Centre, Newport, Isle Of Wight, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fong WCG, Kadalayil L, Lowther S, Grevatt S, Potter S, Tidbury T, Bennett K, Larsson M, Nicolas F, Kurukulaaratchy R, Arshad SH. The efficacy of the Dyson air purifier on asthma control: A single-center, investigator-led, randomized, double-blind, placebo-controlled trial. Ann Allergy Asthma Immunol. 2023 Feb;130(2):199-205.e2. doi: 10.1016/j.anai.2022.10.010. Epub 2022 Oct 23. PMID 36288782
- [Derived] Fong WCG, Grevatt S, Potter S, Tidbury T, Kadalayil L, Bennett K, Larsson M, Nicolas F, Kurukulaaratchy R, Arshad SH. The Efficacy of the Dyson Air Purifier in Improving Asthma Control: Protocol for a Single-Center, Investigator-Led, Randomized, Double-Blind, Placebo-Controlled Trial. JMIR Res Protoc. 2021 Jul 27;10(7):e28624. doi: 10.2196/28624. PMID 34313599

DOCUMENTS (1):
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04729530/ICF_000.pdf